CLINICAL TRIAL: NCT05722600
Title: Effects of Hardaliye, a Fermented Grape Drink, on Oxidative Stress, Lipid Profile and Blood Pressure in Young Footballers: A Randomised Trial
Brief Title: Effects of Hardaliye, a Fermented Grape Drink, on Oxidative Stress, Lipid Profile and Blood Pressure in Young Footballers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ramazan Mert Atan, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RMAtan
Record Dates: First submitted 2023-01-31; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Diet, Healthy; Antioxidative Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hardaliye Group (Experimental): Hardaliye Group consumed 250 ml/day of hardaliye (grape juice) for 28 days.
  Interventions: Other: Grape juice
- Placebo Group (Placebo Comparator): Placebo Group consumed 250 ml/day of placebo drink for 28 days.
  Interventions: Other: Placebo drink

INTERVENTIONS:
Other: Grape juice — Hardaliye (grape juice) is a fermented, traditional non-alcoholic beverage made from fresh grapes. It is mainly produced by the fermentation of grapes, sour cherry leaves and mustard seeds. Hardaliye was purchased from traditional producers in Turkey. Hardaliye Group consumed 250 ml/day of hardaliye (grape juice) for 28 days.
  Arms: Hardaliye Group
Other: Placebo drink — Placebo drink has carbohydrate, energy and sensory properties similar to hardaliye. Placebo Group consumed 250 ml/day of placebo drink
  Arms: Placebo Group

SUMMARY:
In the present study, the authors aimed to investigate the effects of hardaliye (grape juice) consumption on oxidative stress parameters, lipid profile and blood pressure in young football players.

ELIGIBILITY:
Inclusion Criteria:

* Being a male football player playing in a team in the Elite Development League,
* Participating in training with the team at least 5 days a week for 3 months,
* Not consuming red wine, grape juice, and/or hardaliye regularly before the study was started,
* Those who stayed in the sports facility where catering service was provided for breakfast, lunch and dinner were included in the study.

Exclusion Criteria:

* With chronic disease,
* Smoker,
* Those taking antioxidant supplements,
* Non-cooperative subjects or unwilling to sign an informed consent and participate in the study.

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Change in total antioxidant capacity | 28 days
  Measurement of serum level of total antioxidant capacity (μmol Trolox eq/L).
Change in total oxidation status | 28 days
  Measurement of serum level of total oxidation status (μmol H2O2 eq/L).
Change in oxidative stress index | 28 days
  (Serum level of total oxidation status/serum level of total antioxidant capacity) × 100
Change in lipid parameters | 28 days
  Measurement of serum levels total cholesterol (mg/dl), HDL-cholesterol (mg/dl), LDL-cholesterol (mg/dl) and triglycerides (mg/dl).
Change in blood pressure | 28 days
  Measurement of systolic (mm Hg) and diastolic blood pressure (mm Hg)

SECONDARY OUTCOMES:
Change in perceived exercise-induced pain | 28 days
  Perceived exercise-induced pain was determined using the 100-mm Visual Analog Scale. 100-mm Visual Analog Scale scores range from 0 (no pain) to 100 (most severe pain). A higher score indicates a higher perceived pain level.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No